CLINICAL TRIAL: NCT05185388
Title: Socioeconomic Inequalities in the Diagnosis and Treatment of Colon and Ovarian Cancer in England Between 2016-2017: A Data Linkage Study Linking National Cancer Registration and Analysis Service, Hospital Episode Statistics and NHS Digital Datasets
Brief Title: Socioeconomic Inequalities in the Diagnosis and Treatment of Colon and Ovarian Cancer in England Between 2016-2017
Status: Active, not recruiting | Type: Observational
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: RS154-ODR-BPS
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Treatment Related Cancer; Diagnoses Disease; Equality, Gender
Keywords: Socioeconomic Inequalities
MeSH Terms: conditions — Neoplasms, Second Primary; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a population-based, patient-level analysis of colon and ovarian cancer diagnoses in England over a 2-year period using a dataset created by linking NCRAS and NHS digital datasets. Our analyses will look into inequalities in the diagnostic and treatment pathway, and inequalities in treatment received, for those diagnosed with colon and ovarian cancer between 2016-2017.

DETAILED DESCRIPTION:
Colon and ovarian cancer survival in England lags behind other comparable countries. There is also evidence of a deprivation gradient in survival in England, where those from the most deprived areas are more likely to experience a worse survival with the disease.

Inequalities in the diagnostic and treatment pathways, and in treatments received, may contribute to this deprivation gap in survival. This study will look at the secondary care diagnostic interval and the treatment interval to assess for any socioeconomic inequalities in both these intervals. This study will also look at anticancer treatments received (surgery, chemotherapy and the combination of both treatment modalities) to evaluate for any socioeconomic inequalities in treatments received.

Important variables will be adjusted for in statistical modelling, including age, co-morbidities, ethnicity and stage of disease

To evaluate for inequalities in treatments received and diagnostic and treatment intervals the study will use data from the cancer registry, Systemic Anticancer Therapy (SACT), Hospital Episodes Statistics, Diagnostic Imaging Dataset and Cancer Waiting Times datasets. These datasets will be linked by the National Cancer Registration and Analysis Service, using a unique identifier. We will receive a pseudo-anonymised dataset, allowing for patient-level analyses but without identifying individual patients.

ELIGIBILITY:
Inclusion Criteria:

All patients resident in England and aged 18-99 diagnosed with colon cancer (ICD10 C18) or ovarian cancer (ICD10 C48, C56, C57 and D39,1) where the date of diagnosis is between 01/01/2016 and 31/12/2017.

Exclusion Criteria:

Patients with cancers of the appendix (C18.1) will be excluded.

Male patients with ovarian cancer.

Borderline ovarian tumours (ICD-10 site code of C56x, C57x or C48x where the morphology code is: 8442, 8444, 8451, 8463, 8473, 8472 or 8462) and (ICD-10 site code D39.1 where the morphology code is 8144, 8260, 8313, 8380, 8381, 8440, 8441, 8460, 8470, 8480, 8481, 9000, 9013, 9014 or 9015).

Sarcomas are excluded (where the morphology code is: 8693, 8800-8806, 8963, 8990-8991, 9040-9044, 8810, 8811-8921, 9120-9373, 9490, 9500, 9530-9582).

Patients diagnosed with any prior invasive primary malignancies (ICD10 C00-97x), where the date of diagnosis of such prior invasive malignancies precedes the diagnosis date of the first qualifying tumour. Patients with a synchronous diagnosis on the same day as their qualifying tumour will be included within the sample population.

Incomplete registrations excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with colon and ovarian cancer diagnosed between 01/01/2016 and 31/12/2017 in England will be considered for inclusion in the study, according to specific inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 45831 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Inequalities in time to diagnosis and/or treatment | January 2016 - December 2017
  Any differences in time to diagnosis or treatment of colon or ovarian cancer, adjusting for important factors
Inequalities in treatments received | January 2016 - December 2017
  Any differences in treatments received for colon or ovarian cancer, adjusting for important factors

CONTACTS AND LOCATIONS:
Locations (1):
- Hull York Medical School, Hull, Humberside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pickwell-Smith BA, Paton LW, Soyiri I, Lind M, Macleod U. Are there inequalities in ovarian cancer diagnosis and treatment in England? A population-based study. Cancer Epidemiol. 2025 Jun;96:102778. doi: 10.1016/j.canep.2025.102778. Epub 2025 Mar 8. PMID 40058114